CLINICAL TRIAL: NCT00157872
Title: A Multicenter, Randomized, Parallel-Group, 8-Week, Double-Blind, and Active Comparator-Controlled Study to Assess the Efficacy, Safety, and Tolerability of Rofecoxib Tablet 25 mg Once Daily Versus Naproxen Table 500 mg Twice Daily in the Treatment of Chinese Patient With Rheumatoid Arthritis
Brief Title: A Study of Rofecoxib Versus Naproxen in the Treatment of Chinese Patient With Rheumatoid Arthritis (0966-231)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-231; 2005_063
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966; rofecoxib
Drug: Comparator: naproxen tablet 500 mg

SUMMARY:
A study to compare rofecoxib versus naproxen in the treatment of Chinese patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males or females at least 18 years of age with rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-01-07 (Actual); Primary Completion 2004-07-05 (Actual); Study Completion 2004-09-19 (Actual)

PRIMARY OUTCOMES:
Tender joint count
swollen joint count
patient's global assessment of disease activity
investigator's global assessment of disease activity

SECONDARY OUTCOMES:
Patient pain assessment
patient's global assessment of response to therapy
investigator's global assessment of response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html